CLINICAL TRIAL: NCT06468722
Title: Analysis of Fat Oxidation Capacity During Cardiopulmonary Exercise Testing Indicates Long-lasting Metabolic Disturbance in Patients With Post-COVID-19 Syndrome
Brief Title: Fat Oxidation Capacity in Patients With Post Covid-19 Syndrome
Status: Completed | Type: Observational
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Institut für Rehabilitationsforschung Norderney (Unknown)
Responsible Party: Sponsor
Other Study IDs: PCS_Fettoxidation
Record Dates: First submitted 2024-06-19; First posted 2024-06-21 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Post-COVID-19 Syndrome; Long-COVID-19 Syndrome
Keywords: SARS-CoV-2; Long-COVID-19; Exercise-based Rehabilitation; Mitochondrial Dysfunction; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mitochondrial Diseases; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Covid-19 Syndrome Patients
  Interventions: Behavioral: Exercise-based rehabilitation

INTERVENTIONS:
Behavioral: Exercise-based rehabilitation — Patients performed regular physical exercise during inpatient rehabilitation

SUMMARY:
Post-COVID-19 Syndrome (PCS) is characterized by symptoms, including fatigue, reduced physical performance, dyspnea, cognitive impairment, and psychological distress. The mechanisms underlying the onset and severity of PCS point to mitochondrial dysfunction as significant contributor. This study examined fat oxidation as a function of mitochondrial capacity during exercise.

DETAILED DESCRIPTION:
Post-COVID-19 Syndrome (PCS), also known as post-acute sequelae of COVID-19, manifests following an acute infection with the SARS-CoV-2 virus (COVID-19 infection). PCS is characterized by the persistence of symptoms beyond 12 weeks from the onset of infection and/or the emergence of new symptoms within this time. Although recent guidelines offer specific criteria to diagnose PCS, ambiguity persists due to the complex nature of its symptomatology and the lack of definitive diagnostic tools. PCS is a multisystemic disorder characterized by symptoms such as (chronic) fatigue, diminished physical performance, muscular weakness and pain, dyspnea, cognitive impairments and alterations of the autonomous nervous system, as well as mental and psychological distress. The severity of symptoms varies widely among patients, from mild impairment to significant restrictions in daily activities, potentially leading to partial or complete incapacity to work. Of note, the severity of the acute infection does not predict the onset or severity of PCS. Even though many patients experience gradual recovery without specific treatment, there is a substantial need for effective medical rehabilitation, especially for those with persistent PCS. To this respect, exercise-based programs have been shown to induce significantly exercise capacity as well as higher quality of life, reduced fatigue, and less depression. Despite ongoing investigations, the mechanisms contributing to the onset and severity of PCS remain largely unknown. Factors may include endothelial dysfunction and detrimental effects on the microvasculature, as well as a "cytokine storm" associated with excessive oxidative stress and subsequent mitochondrial dysfunction which has emerged as a significant potential contributor.

Notably, detrimental effects on mitochondrial function have been described as a result of severe acute infections triggering an excessive immune response, systemic inflammation and oxidative stress. Recent studies suggested that impaired mitochondrial function in PCS may be associated with impaired fatty acid oxidation (FatOx) which can be identified using cardiopulmonary exercise testing (CPET). Currently, the number of PCS patients characterized for changes in FatOx using CPET is low and associations with signs and symptoms of PCS such as fatigue have not been reported in detail. Moreover, reports on the potential of exercise-based rehabilitation to restore FatOx capacity in PCS are not available. Thus, the current study aimed to investigate if analysis of breath-by-breath spirometric data followed by an estimation of individual FatOx capacity can be used for the stratification of PCS patients. The investigators hypothesized that a lower FatOx potential would be associated with PCS-specific signs and symptoms such as mental and physical fatigue. In addition, the investigators sought to analyze if exercise-based rehabilitation would be effective in restoring PCS patients' FatOx capacity as a sign of improved mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

* a history of (at least one) Covid-19 infection
* ongoing or newly expressed performance deficits lasting for at least 3 months prior to recruitment
* referral to inpatient rehabilitation
* signed informed consent

Exclusion Criteria:

* unstable condition
* incapable of understanding study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Post-COVID-19 syndrome who are referred to Clinic Königsfeld for inpatient medical rehabilitation and who are willing to participate in the study and give their written informed consent. Inclusion criteria were a history of (at least one) COVID-19 infection (positive PCR test at the time of infection), and ongoing or newly expressed performance deficits lasting for at least 3 months prior to recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Change in Fat Oxidation Rate | Baseline and week 4 (i. e. before discharge)
  Fat oxidation will be assessed by breath-by-breath spiroergometry

SECONDARY OUTCOMES:
Change in Carbohydrate Oxidation Rate | Baseline and week 4 (i. e. before discharge)
  Carbohydrate oxidation rate will be assessed by breath-by-breath spirometry
Change in Fatigue | Baseline and week 4 (i. e. before discharge)
  Fatigue will be assessed using the "The Multidimensional Fatigue Inventory (MFI20)"

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic Königsfeld, Ennepetal, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Garbsch R, Schafer H, Mooren FC, Schmitz B. Analysis of fat oxidation capacity during cardiopulmonary exercise testing indicates long-lasting metabolic disturbance in patients with post-covid-19 syndrome. Clin Nutr. 2024 Dec;43(12):26-35. doi: 10.1016/j.clnu.2024.10.010. Epub 2024 Oct 11. PMID 39423759